CLINICAL TRIAL: NCT06184802
Title: Effects of Integrated Therapy Using the Multisensory Room in Autism Spectrum Disorder
Brief Title: Multisensory Room in Autism Spectrum Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Francesca Cucinotta, Principal Investigator, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SENSROOM01
Record Dates: First submitted 2023-12-15; First posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (EG) (Experimental): The group consists of 50 patients diagnosed with autism spectrum disorder, randomly assigned.
  The patients underwent treatment as usual (TAU) integrated with the use of multisensory room, in a 1:1 ratio. All the exercises have been customized by the therapists according to the individual treatment needs, adapting the level of difficulty to the patient's abilities.
  Overall, each patient was treated over a period of 6 months, up to a total of n. 48 sessions, twice a week, lasting 45 minutes each.
  Interventions: Behavioral: TAU+Multisensory room
- Control Group (CG) (Active Comparator): The group consists of 50 patients diagnosed with autism spectrum disorder randomly assigned.
  The patients underwent TAU, consisting in standard neuro-psychomotor training. The treatment was tailored according to each child's goals need and preferences.
  Overall, each patient was treated over a period of 6 months, up to a total of n. 48 sessions, twice a week, lasting 45 minutes each.
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: TAU+Multisensory room — Multisensory room session included exercises in different interaction areas that allow to make up a multisensory experience where the patient can freely perform in different directions experimenting combinations of play
  Arms: Experimental Group (EG)
Behavioral: TAU — neuro-psychomotor training promotes a better organization of global motor skills, improve hand-eye coordination, promote the development of language as communication, enriching representation and symbolization skills.
  Arms: Control Group (CG)

SUMMARY:
Autism spectrum disorder (ASD) is a complex neurological development with onset in infancy or early childhood. Atypical sensory processing has been widely reported in ASD, and recent literature suggest that this abnormality extends across the life span, with consequent important implications in every-day life of autistic individuals and their families. Multisensory environments have been used in children with ASD precisely as a function of this particular difference in sensory processing and some studies have highlighted potential benefits. Therefore, the aim of our study is to verify feasibility and efficacy of an integrated treatment program with the multisensory room compared to as usual treatment in patients with ASD.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a complex neurological development with onset in infancy or early childhood. In the Fifth Edition of Diagnostic and Statistical Manual of Mental Disorders, sensory features were finally take into account and atypical responses to sensory stimuli was included in the diagnostic criterion, such as the presence of hyper- or hypo-responsiveness to sensory inputs or unusual interests towards sensory aspects of the environment, and it must be considered (APA 2013). Atypical sensory processing has been widely reported in ASD, and recent literature suggest that this abnormality extends across the life span, with consequent important implications in every-day life of autistic individuals and their families.

Multisensory environments have been used in children with ASD precisely as a function of this particular difference in sensory processing and some studies have highlighted potential benefits. The multisensory rooms were designed to provide multiple stimulation opportunities that cover all sensory channels. Among the present literature data, interventions targeting sensory integration seems to be useful in reducing challenging behaviors in many individuals with developmental disabilities including ASD (Novakovic N. et al. 2019; Kaplan H. et al., 2006; McKee et al. 2007). The aim of our study is to verify feasibility and efficacy of an integrated treatment program with the multisensory room compared to as usual treatment in patients with ASD.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with diagnosis of ASD, according to Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria;
* age between 3 and 6 years;
* signed informed consent and the availability of at least one family member to participate in the diagnostic/therapeutic process.

Exclusion Criteria:

* children not aged between 3 and 6 years;
* significant medical conditions such as epilepsy, significant visual and auditory sensory deficits, traumatic brain injury, or significant genetic disorders.
* Informed consent not signed of at least one family member to participate in the diagnostic/therapeutic process.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2019-11-04 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Psychoeducational Profile, Third Edition (PEP-3) | T0 (Baseline) - T1 (6 Months)
  a scale to assess developmental skills and behaviors of children with autism and communication disabilities, aged between 6 months and 7 years. It identifies learning strengths and emerging abilities concerning communication, motor skills and maladaptive behaviors
Childhood Autism Rating Scale (CARS-2) | T0 (Baseline) - T1 (6 Months)
  The CARS 2 evaluates the child's behavior in several areas, including verbal and nonverbal communication, socialization, stereotyped and repetitive behavior, and adaptation to change. It is made up of 15 questions with a rating scale ranging from 1 to 4, where 1 indicates normal behavior and 4 indicates highly anomalous behavior. It is possible to obtain a score between 15 and 60, where a higher score indicates a greater severity of ASD symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Neurolesi Bonino Pulejo, Messina, Italy

REFERENCES:
- [Background] Novakovic N, Milovancevic MP, Dejanovic SD, Aleksic B. Effects of Snoezelen-Multisensory environment on CARS scale in adolescents and adults with autism spectrum disorder. Res Dev Disabil. 2019 Jun;89:51-58. doi: 10.1016/j.ridd.2019.03.007. Epub 2019 Mar 29. PMID 30933867
- [Background] Kaplan H, Clopton M, Kaplan M, Messbauer L, McPherson K. Snoezelen multi-sensory environments: task engagement and generalization. Res Dev Disabil. 2006 Jul-Aug;27(4):443-55. doi: 10.1016/j.ridd.2005.05.007. Epub 2005 Aug 24. PMID 16122905
- [Background] McKee SA, Harris GT, Rice ME, Silk L. Effects of a Snoezelen room on the behavior of three autistic clients. Res Dev Disabil. 2007 May-Jun;28(3):304-16. doi: 10.1016/j.ridd.2006.04.001. Epub 2006 Jun 27. PMID 16806812
- [Background] American Psychiatric Association. (2013). Diagnostic and statistical manual of mental disorders (DSM-5®). Biobehavioral Reviews, 33, 1204-1214